CLINICAL TRIAL: NCT02433730
Title: The Effect of Testosterone Replacement in Patients With Hypogonadotrophic Hypogonadism Due to Opioid Treatment for Non-malignant Disease
Brief Title: Testosterone Therapy in Hypogonadal Men Treated With Opioids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marianne Andersen (Other)
Responsible Party: Sponsor-Investigator, Marianne Andersen, Professor, MD,, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22102014
Record Dates: First submitted 2015-01-27; First posted 2015-05-05 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Active Comparator): intramuscular injection
  Interventions: Drug: placebo
- testosterone (Active Comparator): intramuscular injection
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — intramuscular injection
  Other Names: nebido
  Arms: testosterone
Drug: placebo — intramuscular injection
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of testosterone replacement therapy in men with low testosterone due to opioid treatment on body composition, the haemostatic system, glucose metabolism, muscle function, pain sensitivity, pain modulation, lipids, sexual function and quality of life.

Male patients on opioids for non-malignant diseases aged 18-59 years diagnosed with hypogonadotrophic hypogonadism, referred from day hospitals and outpatient populations. 40 patients are randomized to either testosterone undecanoate i.m. or placebo i.m., i.e. 20 patients per arm

A double blinded randomized placebo controlled trial

DETAILED DESCRIPTION:
The study duration is 24 weeks. Patients are treated with Testosterone Undecanoate 1000 mg/4 ml, intramuscular (i.m.) or placebo at 0, 6 and 18 weeks.

Outcome measures will be evaluated at 0 and 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18-75 years
* Treatment with opioid for >3 months, daily dose >50-100 mg
* Total testosterone < 12 mmol/L
* Follicle Stimulating Hormone (FSH)/Luteinizing Hormone (LH) levels normal og below normal laboratory values
* Normal prolactin levels

Exclusion Criteria:

* Hematocrit> 54% at screening
* Prostate Specific Antigen (PSA) > 3 ng/ml
* Severe organic and mental disease
* current or present cancer diagnosis
* Previous venous thrombotic embolism and cerebrovascular disease
* Uncontrolled hypertension
* Epilepsy or migraine not adequately controlled by therapy
* Severe benign prostate hypertrophy with symptom score >19
* Sleep apnea
* Alcohol or drug abuse
* Implantation of sustained action sex hormone in the last 12 months
* Use of oral, buccal or transdermal testosterone in the last two weeks
* Treatment with glucocorticoids > 5 mg/day or 5 alfa reductase inhibitors
* Hypersensitivity to Nebido

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
lean body mass | 24 weeks
  dual xray absorptiometry scan

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odensen, Denmark

REFERENCES:
- [Derived] Olesen TB, Glintborg D, Johnk F, Olsen MH, Andersen MS. Blood pressure responses to testosterone therapy are amplified by hematocrit levels in opioid-induced androgen deficiency: a double-blind, randomized, placebo-controlled trial. J Hypertens. 2024 May 1;42(5):893-901. doi: 10.1097/HJH.0000000000003638. Epub 2023 Dec 13. PMID 38088425